CLINICAL TRIAL: NCT04104984
Title: Antenatal Management Based on Transvaginal Ultrasound Cervical Length Screening for Preventing Preterm Birth
Brief Title: Detection of Preterm Labour by Cervical Length
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shehab Alam Millad, principle investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VUS cervical Length
Record Dates: First submitted 2019-09-17; First posted 2019-09-26 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-09

CONDITIONS: Preterm Labour
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Tocolytic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group not follow NICE guide lines (Experimental): All pregnant women who fulfil the same inclusion criteria, exclusion criteria, diagnoses established as short cervix , and do not managed according to NICE guide lines will be treated and managed according to their units as a control group.
  Interventions: Other: digital vaginal exam; Device: abdominal ultrasound; Drug: Tocolytic Agents
- study group follow NICE guide lines (Experimental): - All pregnant women will attend hospital between 14-24 weeks and fulfil inclusion and exclusion criteria will be approached for possibility to be included in the study . and will be managed according NICE guide lines
  Interventions: Device: transvaginal ultrasound; Drug: Progesterone Vaginal Suppository; Procedure: cervical cercalage

INTERVENTIONS:
Device: transvaginal ultrasound — a transvaginal ultrasound is done to patient to determine cervical length
  Arms: study group follow NICE guide lines
Drug: Progesterone Vaginal Suppository — a progesterone vaginal suppository to prevent preterm labour
  Arms: study group follow NICE guide lines
Procedure: cervical cercalage — Mcdonald's cervical cercalage . a stitch taken around the cervix to prevent preterm labour
  Arms: study group follow NICE guide lines
Other: digital vaginal exam — vaginal examination to detect short cervix
  Arms: control group not follow NICE guide lines
Device: abdominal ultrasound — use abdominal ultrasound to measure cervical length
  Arms: control group not follow NICE guide lines
Drug: Tocolytic Agents — a medication is given to prevent uterine contraction
  Arms: control group not follow NICE guide lines

SUMMARY:
Detection of short cervix by transvaginal ultrasound and its evidence based management to prevent preterm birth .

DETAILED DESCRIPTION:
* All pregnant women will attend hospital between 14-24 weeks and fulfil inclusion and exclusion criteria will be approached for possibility to be included in the study .
* History taking .Obstetric history will be obtained from the patient includes gravidity and parity , last menstrual period , duration of gestation at birth time , mode of delivery , gender, birth Wight, any complication in each pregnancy, miscarriage and causes of miscarriage . Past history will be obtained from the patient for any medical disease like ( severe anaemia, hypertensive disease, heart disease, antiretroviral therapy in pregnancy and genitourinary infection) and History of cervical cercalage . Family history will be obtained to determine any history of family preterm birth. Socioeconomic status will be obtained include occupation and financial status. Special Habits for both couples.

  * Gynaecological history will be taken from the patient include any vaginal bleeding, history of vaginal infection, operations like D and C with cervical dilatation.
  * Examination Examination of the patient include vital signs, general examination ( head, neck ,chest ,heart ) obstetric examination include inspection, palpation, auscultation and speculum vaginal examination.
  * -Investigation Investigation includes antenatal care laboratory tests like urine analysis ,CBC, RH factor and random blood sugar .
  * Transvaginal ultrasound:

Study group : Cervical length will be measured using transvaginal ultrasonography with the standard longitudinal view of cervix while patient's bladder is empty. TVS probe will be used to measure cervical length. It will be measured by keeping the probe 3cm away from the posterior fornix. The cervical length is defined as the length between the internal OS and external OS

Those with short cervix less than 25 mm will be managed According to NICE guide lines :

Offer a choice of either prophylactic vaginal progesterone or prophylactic cervical cerclage to women: with a history of spontaneous preterm birth or mid-trimester loss between 16+0 and 34+0 weeks of pregnancy and in whom a transvaginal ultrasound scan has been carried out between 16+0 and 24+0 weeks of pregnancy that reveals a cervical length of less than 25 mm.

Discuss the benefits and risks of prophylactic progesterone and cervical cerclage with the woman and take her preferences into account.

Offer prophylactic vaginal progesterone to women with no history of spontaneous preterm birth or mid-trimester loss in whom a transvaginal ultrasound scan has been carried out between 16+0 and 24+0 weeks of pregnancy that reveals a cervical length of less than 25 mm.

Consider prophylactic cervical cerclage for women in whom a transvaginal ultrasound scan has been carried out between 16+0 and 24+0 weeks of pregnancy that reveals a cervical length of less than 25 mm and who have either: had preterm prelabour rupture of membranes (P-PROM) in a previous pregnancy or a history of cervical trauma (17) .

progesterone will be given in form of vaginal suppository 200 mg once daily . Start receiving it once diagnoses is established till 34 week gestation.

A McDonald cerclage will be be preformed for women once diagnoses is established and removed at 36 week gestational or when labour pain start.

Control group : All pregnant women who fulfil the same inclusion criteria, exclusion criteria, diagnoses established as short cervix by digital vaginal exam or trans abdominal ultrasound or not specified and do not undergo transvaginal ultrasound assessment , and do not managed according to NICE guide lines will be treated and managed according to their units as a control group.

• Then all patients will be followed up every 4 weeks by taking history , any complaint of new symptoms , compliance to treatment, obstetric exam and investigation if indicated till delivery and record the time of delivery or termination of pregnancy. After delivery, record maternal and fetal outcome.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gestational age between 14-24 weeks and having singletone or multiple viable fetus

Exclusion Criteria:

.Current Cervical cercalage.

* Major Fetal malformation .
* Prenatal infection (bacterial vaginosis ) .Medical comorbidities . .Currently receiving Progesterone treatment. .Pregnancy from assisted reproductive technique . .Threatened miscarriage . .Rupture membrane. .Painful uterine contraction. .Low implanted placenta.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 966 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
preterm birth, defined as delivery before 37 weeks 0 days of gestation | baseline
  determine number of patients with preterm birth under 37 week gastational age and trying to prevent early diagnosed conditions from 922 patient diagnosed with short cervix

SECONDARY OUTCOMES:
Mean GA at delivery | baseline
  detection of Mean gastational age at delivery
Birth Wight less than 2500 grams. | baseline
  determine number of infants born from patients with short cervix and undergo management and record Birth Wight less than 2500 grams.
Birth Wight ( mean +SD) in grams | baseline
  detection of Birth Wight ( mean +SD) in grams
compliance to medication. | baseline
  determine if the 466 of study group patient taking the medication regularly as progesterone vaginal suppository by questioning the patient.
side effect related to intervention either progesterone or cercalage | baseline
  detection and record the side effect related to intervention either progesterone or cercalage by questioning the patient
Mode of delivery | baseline
  recording which patients deliver normal vaginal delivery or by cesarean section
perinatal mortality. | baseline
  record the numbers of perinatal death who's mothers undergo treatment during pregnancy of overall 922 patients
Neonatal morbidity | baseline
  record infants born to mother of study group and study group after birth with any morbidity like respiratory distress syndrome,necrotizing enterocolities,jaundice .
admission to Neonatal intensive care unit | baseline
  determine which infant born will be admitted to the intensive care unit after delivery and record numbers of infants .
Maternal morbidity | baseline
  record Maternal morbidity like maternal haemorrhage , maternal infection ,maternal medication from 922 patients with short cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Eldeen M Ismail, MD, Principal Investigator — Asssiut University; Ahmed M Alaa eldeen, MD, Principal Investigator — Assiut University; Hany A Ali, MD, Principal Investigator — Asssiut University